CLINICAL TRIAL: NCT06628596
Title: Acute Effects of Paraxanthine on Energy, Focus, Appetite, and Cognition: Double-Blind, Placebo-Controlled Trial
Brief Title: Acute Effects of Paraxanthine on Energy and Focus
Acronym: PXN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Iovate Health Sciences International Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IOV-001-032024
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Cognition; Appetite; Mental Energy; Dietary Supplement
Keywords: cognition; appetite; mental energy; mental focus; dietary supplement
MeSH Terms: interventions — 1,7-dimethylxanthine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): After qualifying for the study, subjects will be randomly assigned to receive a placebo, 200mg PXN, and 300mg PXN using a Latin Square design.
  * Paraxanthine (200 mg)
  * Paraxanthine (300 mg)
  * Placebo (containing 300mg resistant starch) •Supplements will be provided in identical-looking capsules with label directions and Study Protocol Number.
  Interventions: Dietary Supplement: Paraxanthine 200mg and 300mg
- Paraxanthine 200mg (Active Comparator): After qualifying for the study, subjects will be randomly assigned to receive a placebo, 200mg PXN, and 300mg PXN using a Latin Square design.
  * Paraxanthine (200 mg)
  * Paraxanthine (300 mg)
  * Placebo (containing 300mg resistant starch) •Supplements will be provided in identical-looking capsules with label directions and Study Protocol Number.
  Interventions: Dietary Supplement: Paraxanthine 200mg and 300mg
- Paraxanthine 300mg (Active Comparator): After qualifying for the study, subjects will be randomly assigned to receive a placebo, 200mg PXN, and 300mg PXN using a Latin Square design.
  * Paraxanthine (200 mg)
  * Paraxanthine (300 mg)
  * Placebo (containing 300mg resistant starch) •Supplements will be provided in identical-looking capsules with label directions and Study Protocol Number.
  Interventions: Dietary Supplement: Paraxanthine 200mg and 300mg

INTERVENTIONS:
Dietary Supplement: Paraxanthine 200mg and 300mg — Participants consumed 200 mg paraxanthine (PXN 200), 300 mg paraxanthine (PXN 300), or placebo (PLA) after an overnight fast. Supplements were ingested 30 minutes before a mixed meal in double-blind, randomized, placebo-controlled, crossover fashion.
  Other Names: Placebo (PLA); Paraxanthine 200mg (PXN 200); Paraxanthine 300mg (PXN 300)

SUMMARY:
This study aims to evaluate the effects of paraxanthine (200 mg and 300 mg) on energy, focus, appetite, and cognitive performance in healthy adults. Using a double-blind, placebo-controlled, crossover design, participants will receive paraxanthine or placebo 30 minutes before a meal. Cognition tests and visual Analogue Scale (VAS) ratings for energy, focus, productivity, satiety, and appetite will be collected at multiple time points post-consumption.

DETAILED DESCRIPTION:
Caffeine (CAF) is one of the most consumed naturally occurring nootropic and exercise-related ergogenic aids. Paraxanthine (1,7-dimethylxanthine, PXN) is the main metabolite of CAF, accounting for 70-72% of CAF ingested, and 85% of the methylxanthine metabolic by-products. While caffeine has been extensively studied for its effects on energy, and focus in humans, the effects of paraxanthine are less understood.

It was recently reported that acute ingestion of PXN enhances various markers of focus such as memory, reaction time, and attention for up to 6-hours in healthy adults, and that acute ingestion as low as 50 mg of PXN for 7-days enhanced measures of cognition, memory, reasoning, response time, and helped sustain attention. While studies were performed in the fasted state and over 6 hours which is beyond the ~3.1h half-life of paraxanthine, the cognitive effects of paraxanthine in response to an ecologically valid meal over a 3-hour period is limited. Therefore, the purpose of this study is to assess the impact of paraxanthine on energy, focus, and cognition in younger healthy adults in the fed state.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily provide signed and dated informed consent.
* Be in good health as determined by medical history and routine blood chemistries.
* Age between 20 and 40 years (inclusive).
* Body Mass Index of 18.5-29.9 (inclusive).
* Body weight of at least 120 pounds.
* Normotensive (supine, resting systolic blood pressure <140 mm Hg and diastolic blood pressure < 90 mm Hg. If the first measurement is slightly elevated above these limits, the subject will be given a brief (5 minute) rest period, and two more measurements will be taken. The average of all three measurements will be used to determine eligibility.
* Normal supine, resting heart rate (< 90 per minute).
* Willing to duplicate their previous 24-hour diet, refrain from alcohol, caffeine, and exercise for 24 hr prior to each trial, and fast for 8 hours prior to each trial.

Exclusion Criteria:

* Current smoker or other nicotine use (i.e. vape, patch, etc.).
* History of malignancy in the previous 5 years except for non-melanoma skin cancer (basal cell cancer or squamous cell cancer of the skin).
* Prior gastrointestinal bypass surgery (Lapband, etc.).
* Other known gastrointestinal or metabolic diseases that might impact nutrient absorption or metabolism, e.g. electrolyte abnormalities, diabetes, thyroid disease, adrenal disease, hypogonadism, short bowel syndrome, diarrheal illnesses, history of colon resection, gastric ulcer, reflux disease, gastroparesis, Inborn-Errors-of-Metabolism (such as PKU).
* Chronic inflammatory condition or disease (e.g. rheumatoid arthritis, Crohn's disease, ulcerative colitis, Lupus, HIV/AIDS, etc.).
* History of hepatorenal, musculoskeletal, autoimmune, or neurologic disease.
* History of cognitive disorder.
* History of psychiatric disorder.
* Known sensitivity to any ingredient in the test formulations as listed in the Certificates-of-Analysis.
* Women currently pregnant, trying to become pregnant or breastfeeding a child.
* Use of anxiety or ADHD medication.
* Caffeine intake of three or more cups of coffee or equivalent (>400 mg) per day.
* Alcohol consumption (more than 2 standard alcoholic drinks per day or more than 10 drinks per week) or drug abuse or dependence.
* Clinically significant abnormal laboratory results at screening.
* Prior gastrointestinal bypass surgery (Lapband, etc.).
* Currently participating in another research study with an investigational product or have been in another research study in the past 30 days.
* Any other diseases or conditions that, in the opinion of the medical staff, could confound the primary endpoint or place the subject at increased risk of harm if they were to participate.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biological males and females.
Enrollment: 25 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Energy | Energy (via visual analogue scale) measured at -30, 0 (meal), and 30, 60, 120, 180 minutes post-meal.
  Using 100 mm anchored visual analogue scale. Higher scores indicate an improvement.
Focus | Focus (via visual analogue scale) measured at -30, 0 (meal), and 30, 60, 120, 180 minutes post-meal.
  Using 100 mm anchored visual analogue scale. Higher scores indicate an improvement.
N-Back Task | Assessed at t = - 30min (prior to study product ingestion) and at t = 0 min immediately before the standardized mealand 30-, 60-, 120-, and 180 minutes post meal ingestion.
  Two repetitions of the N-Back Task (90s in duration) to assess memory, attention and decision making
Go/No-Go Task | Assessed at t = - 30min (prior to study product ingestion) and at t = 0 min immediately before the standardized mealand 30-, 60-, 120-, and 180 minutes post meal ingestion.
  Two repetitions of the Go/No-Go Task (90s in duration) to assess measures of attention, processing speed and impulse control
Serial 7s | Assessed at t = - 30min (prior to study product ingestion) and at t = 0 min immediately before the standardized mealand 30-, 60-, 120-, and 180 minutes post meal ingestion.
  Two repetitions of Serial 7s (90s in duration) to assess attention, working memory, and mental arithmetic's.

SECONDARY OUTCOMES:
Satiety/Feelings of fullness | Satiety/Feelings of fullness (via visual analogue scale) measured at -30, 0 (meal), and 30, 60, 120, 180 minutes post-meal.
  Using 100 mm anchored visual analogue scale. Higher scores indicate an improvement.
Appetite | Appetite (via visual analogue scale) measured at -30, 0 (meal), and 30, 60, 120, 180 minutes post-meal.
  Using 100 mm anchored visual analogue scale. Higher scores indicate an improvement.
Productivity | Productivity (via visual analogue scale) measured at -30, 0 (meal), and 30, 60, 120, 180 minutes post-meal.
  Using 100 mm anchored visual analogue scale. Higher scores indicate an improvement.

OTHER OUTCOMES:
Safety (vital signs, side effect profile/AE monitoring). | Over the 3.5 hour measurement period
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- The Center For Applied Health Sciences, Canfield, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
Case by case basis.

REFERENCES:
- See also: The Center For Applied Health Sciences Website — https://thecahs.com/current-studies